CLINICAL TRIAL: NCT06966310
Title: Awake Prone Positioning of Patients Suffering Community Acquired Pneumonia Requiring Nasal High Flow Therapy, Excluding COVID-19
Brief Title: Awake Prone Positioning of Patients Suffering Community Acquired Pneumonia Requiring Nasal High Flow Therapy
Acronym: PRONECAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR230003
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone position group (Experimental): patients will be invited and assisted to prone as long as possible every day. The goal is to achieve at least 8h in the prone position per 24h period, with 3-6 prone sessions.
  Interventions: Other: Prone position
- Control group (No Intervention): Usual care including nasal high flow therapy adapted for a SpO2 of 92-95%. No prone positioning.

INTERVENTIONS:
Other: Prone position — depending on tolerance, the objective is to spend as much time as possible, up to 16h and beyond, in prone position per period of 24 hours. For each session the patients will be encouraged to stay as long as possible in the prone position (i.e. ideally 4-8 hours each session).
  Arms: Prone position group

SUMMARY:
Community acquired pneumonia, in particular when requiring oxygen therapy because of acute hypoxemic respiratory failure and meeting acute respiratory distress syndrome (ARDS) criteria frequently leads to tracheal intubation and poor outcome.

Among invasively mechanically ventilated patients with ARDS and presenting a PaO2/FiO2 ratio (arterial partial pressure of oxygen to inspired fraction of oxygen) of less than 150 mmHg, the prone position significantly reduces mortality and represents standard care (Guérin 2013). Among non-intubated COVID-19 patients, a subtype of viral community acquired pneumonia, a recent study showed that awake prone positioning reduces the composite outcome of intubation or death among patients requiring nasal high flow therapy. Furthermore, it favored weaning of nasal high flow therapy.

Prone position in patients with non-COVID ARDS treated with high nasal flow was evaluated in 20 patients with predominantly viral pneumonia (Ding 2020) and was associated with improved oxygenation.

We hypothesize that prone positioning of patients suffering non-COVID community acquired pneumonia and undergoing nasal high flow therapy can significantly improve outcome by reducing the need for intubation and associated therapies such as sedation and muscle relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to an intensive care unit or intermediate care unit
* Suspicion of community acquired pneumonia (at least one of the 3 criteria): fever, cough, purulent expectoration
* And abnormalities suggestive of pneumonia by chest X-ray or CT-scan
* PaO2/FiO2 ratio <300 mmHg (or equivalent SpO2/FiO2 i.e. < 315 mmHg) under a minimum gas flow of 30 L/min.
* Person affiliated to a French social security system or equivalent
* Informed consent.

Exclusion Criteria:

* Positive SARS-COV2 test within the last 30 days
* Indication for immediate intubation
* Patients for whom a "do not intubate" decision has been made
* Chest trauma or other contraindication to prone position
* Patients with formal indication for non-invasive ventilation: exacerbation of chronic obstructive pulmonary disease, acute cardiogenic pulmonary oedema.
* Pregnant or breastfeeding woman
* Subjects who are under legal protection measure
* More than 8h awake prone positioning prior to inclusion
* More than 48h since intensive care unit or intermediate care unit admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1078 (Estimated)
Dates: Start 2025-05-19 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Intubation within 28 days of randomization | From randomization to day 28
  Analyzed in a competing risk framework with death and intensive care unit discharge taken into account as competing events.

SECONDARY OUTCOMES:
Patient comfort before the first prone session, using a visual analogue scale. | From randomization to 6 hours
Patient comfort during the first prone session, using a visual analogue scale. | From randomization to day 1
Patient comfort after the first prone session, using a visual analogue scale. | From randomization to day 1
Oxygenation (PaO2/FiO2 ratio and ROX index [ratio of SpO2/FiO2 to respiratory rate, Roca 2019]) before the first prone session for patients in the intervention group. | From randomization to 6 hours
Oxygenation (PaO2/FiO2 ratio and ROX index [ratio of SpO2/FiO2 to respiratory rate, Roca 2019]) during the first prone session for patients in the intervention group. | From randomization to day 1
Oxygenation (PaO2/FiO2 ratio and ROX index [ratio of SpO2/FiO2 to respiratory rate, Roca 2019]) after the first prone session for patients in the intervention group. | From randomization to day 1
Daily patient comfort comparison between groups from day 1 to day 3, using a visual analogue scale. | From day 1 to day 3
Oxygenation (PaO2/FiO2 ratio and ROX index) daily comparison between groups from day 1 to day 3. | From day 1 to day 3
Time to treatment escalation to non-invasive ventilation or continuous positive airway pressure (CPAP) with intubation or death as competing events (up to day 28 or intensive care unit discharge whichever occurs first). | From randomization to day 28 or intensive care unit discharge whichever occurs first
Time to successful weaning of nasal high flow with intubation or death as competing events (up to day 28 or intensive care unit discharge whichever occurs first). | From randomization to day 28 or intensive care unit discharge whichever occurs first
Time to intensive care unit discharge and time to hospital discharge (up to day 28). | From randomization to day 28
Mortality | From randomization to day 90
Mortality | From randomization to day 28 or intensive care unit and hospital discharge
Nursing workload: time spent in the patient room by nursing staff during the 24 hours post randomization in both groups | From randomization to 24 hours post randomization
  measured as person.hours
Evolution of patient's quality of life | At 90 days
  using the EQ-5D-5L questionnaire
Evolution of patient's quality of life | At 5 years
  using the EQ-5D-5L questionnaire
Safety: skin lesions, lines dislodgement, central line infection, vomiting, (up to day 28 or intensive care unit discharge whichever occurs first). | From randomization to day 28 or intensive care unit discharge whichever occurs first).

CONTACTS AND LOCATIONS:
Overall Officials: Stephan EHRMANN, Study Director — University Hospital, Tours
Locations (35):
- France (35):
  - Intensive care, University Hospital, Amiens, Amiens
  - Intensive care, University Hospital, Angers, Angers
  - Intensive care, University Hospital, Argenteuil, Argenteuil
  - Intensive care, University Hospital, Belfort, Belfort
  - Intensive care, University Hospital, Besancon, Besançon
  - Intensive care, University Hospital, Bethune, Béthune
  - Intensive care, University Hospital, Blois, Blois
  - Intensive care, University Hospital, Bordeaux, Bordeaux
  - Intensive care, University Hospital, Bourg en Bresse, Bourg-en-Bresse
  - Intensive care, University Hospital, Bourges, Bourges
  - Intensive care, University Hospital, Brest, Brest
  - Intensive care, University Hospital, Colombes, Colombes
  - Intensive care, University Hospital, Dieppe, Dieppe
  - Intensive care, University Hospital, Dijon, Dijon
  - Intensive care, University Hospital, Dreux, Dreux
  - Intensive care, University Hospital, Garches, Garche
  - Intensive care, University Hospital, Grenoble, Grenoble
  - Intensive care, University Hospital, La Roche sur Yon, La Roche-sur-Yon
  - Intensive care, University Hospital, Le Mans, Le Mans
  - Intensive care, University Hospital, Lens, Lens
  - Intensive care, University Hospital, Lille, Lille
  - Intensive care, University Hospital, Lorient, Lorient
  - Intensive care, University Hospital, Lyon, Lyon
  - Intensive care, University Hospital, Morlaix, Morlaix
  - Intensive care, University Hospital, Nantes, Nantes
  - Intensive care, University Hospital, Nice, Nice
  - Intensive care, University Hospital, Orléans, Orléans
  - Intensive care, University Hospital, Cochin, Paris
  - Intensive care, University Hospital, Tenon, Paris
  - Intensive care, University Hospital, Poitiers, Poitiers
  - Intensive care, University Hospital, Rouen, Rouen
  - Intensive care, University Hospital, Saint Brieuc, Saint-Brieuc
  - Intensive care, University Hospital, Saint Nazaire, Saint-Nazaire
  - Intensive care, University Hospital, Strasbourg, Strasbourg
  - Intensive care, University Hospital, Tours, Tours